CLINICAL TRIAL: NCT03130530
Title: Retrospective Study on Colorectal Robotic Surgery Results Obtained Using a New Robotic Platform
Status: Completed | Type: Observational
Sponsor: Istituto Clinico Humanitas (Other)
Responsible Party: Sponsor
Other Study IDs: RETROSPECTIVE-2016
Record Dates: First submitted 2017-04-19; First posted 2017-04-26 (Actual); Last update posted 2017-04-26 (Actual); Status verified 2017-04

CONDITIONS: Colorectal Surgery
Keywords: robotic; colorectal; surgery

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- ALF-X: all patient underwent robotic colorectal surgery using ALF-X system

SUMMARY:
The ALF-X (Advanced Laparoscopy through Force reflection) Robotic Surgery System is a medical device that is available for distribution in the EU (European Union) under CE Mark for use in general surgery, thoracic surgery, gynecological surgery and urological surgery. The main research question is to assess, from a retrospective poit of view, the safety and feasibility of this new robotic platform in the colorectal surgery.

DETAILED DESCRIPTION:
The rationale of this study is to investigate the perioperative and the short term perioperative outcomes of this new robotic Platform in minimally invasive colorectal surgery. Tha ALF-X utilizes fully reusable along with haptic feedback and an innovative vision control system.

ELIGIBILITY:
Inclusion Criteria:

* Patients affected by colorectal disease (benign or malignant) having undergone surgery using ALF-X platform

Exclusion Criteria:

* none

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients indicated for colorectal surgery using ALF-X Robotic surgery system
Sampling Method: Non-Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2015-06-01 (Actual); Primary Completion 2016-09-30 (Actual); Study Completion 2016-09-30 (Actual)

PRIMARY OUTCOMES:
Evaluation adverse events | from the surgery up to 30 days after the surgery
  Adverse events occurred during the surgery and during the 30 days after the surgery evaluated using Clavien-Dindo Classification, conversion rate to traditional laparoscopy or open surgery

SECONDARY OUTCOMES:
Duration of hospitalisation | from surgery to hospital discharge, up to 30 days
  Duration of hospitalisation
Duration of surgery | from to the start to the end of the surgery
  Duration of surgery
Setup for surgery - collision rate | from to the start to the end of the surgery
  Registration and calculation of the collision rate
Setup for surgery - reduced mobility | from to the start to the end of the surgery
  Registration and calculation of the reduced mobility of the tools
Adverse events | Up to 30 days post-surgery
  Number of adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Antonino Spinelli, Prof., Principal Investigator — Istituto Clinico Humanitas

IPD SHARING:
Plan to Share IPD: No